CLINICAL TRIAL: NCT02532764
Title: Phase 1b, Randomized, Double-blind, Placebo-controlled, Dose Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of QR-010 in Subjects With Homozygous ΔF508 Cystic Fibrosis
Brief Title: Dose Escalation Study of QR-010 in Homozygous ΔF508 Cystic Fibrosis Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ProQR Therapeutics (Industry)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: PQ-010-001
Record Dates: First submitted 2015-08-13; First posted 2015-08-26 (Estimated); Results first posted 2019-02-06 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-01

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; ΔF508; RNA therapies; antisense oligonucleotide; CFTR; F508del; CF; RNA therapy
MeSH Terms: conditions — Cystic Fibrosis | interventions — eluforsen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- QR-010 (Experimental): QR-010 administered via inhalation either as a single dose or three times weekly for four weeks.
  Interventions: Drug: QR-010
- Placebo (Placebo Comparator): Placebo (normal saline) administered via inhalation either as a single dose or three times weekly for four weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QR-010 — Single-stranded RNA antisense oligonucleotide in aqueous solution for oral inhalaton
  Arms: QR-010
Drug: Placebo — Normal Saline
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled study of single and multiple ascending doses of QR-010 in adults homozygous for ΔF508 Cystic Fibrosis.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety, tolerability, and to determine the pharmacokinetics of QR-010 administered via inhalation in adult homozygous for ΔF508 Cystic Fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CF as defined by iontophoretic pilocarpine sweat chloride test (sweat chloride) of > 60 mmol/L
* Confirmation of CFTR gene mutations homozygous for the ΔF508 mutation
* Body mass index (BMI) ≥ 17 kg/m2
* Non-smoking for a minimum of two years
* FEV1 ≥70% of predicted normal for age, gender, and height, at Screening
* Stable lung function
* Adequate hepatic and renal function

Exclusion Criteria:

* Breast-feeding or pregnant
* Use of lumacaftor or ivacaftor
* Use of any investigational drug or device
* History of lung transplantation
* Hemoptysis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2015-06; Primary Completion 2017-09-14 (Actual); Study Completion 2017-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Elborn, MD, Principal Investigator — Trust and Queen's University Belfast
Locations (27):
- United States (12):
  - University of Southern California USC - Keck School of Medicine, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Northwestern University, Chicago, Illinois
  - University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Washington Medical Center, Seattle, Washington
- Belgium (2):
  - Universitair Ziekenhuis Brussel, Brussels
  - University of Leuven, Leuven
- University of Calgary (Health Sciences Centre), Calgary, Alberta, Canada
- Motol University Hospital, Prague, Czechia
- Cystic Fibrosis Center Rigshospitalet, Copenhagen, Denmark
- France (2):
  - HGRL Chu Nantes, Nantes
  - Hopital Necker- Enfants Malades, Paris
- Germany (3):
  - Charité Universitätsmedizin Berlin, Berlin
  - Medizinische Hochschule Hannover, Hanover
  - Munich U. Hospital, Cystic Fibrosis Center for Adults, Munich
- Azienda Ospedaliera Universitaria Integrata di Verona, Verona, Italy
- Hospital Vall D'Hebron, Barcelona, Spain
- United Kingdom (3):
  - Celerion, Belfast, Northern Ireland
  - Royal Brompton Hospital, London
  - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Miah KM, Hyde SC, Gill DR. Emerging gene therapies for cystic fibrosis. Expert Rev Respir Med. 2019 Aug;13(8):709-725. doi: 10.1080/17476348.2019.1634547. Epub 2019 Jun 27. PMID 31215818

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment of this clinical trial followed a staggered approach; a new SAD cohort was enrolled following review of the previous SAD cohort. The first MAD cohort opened following the review of the first two SAD cohorts. Subsequent MAD dosing cohorts were initiated following review of the corresponding supportive SAD and MAD cohorts.
Groups:
- QR-010 SAD 6.25mg; QR-010 SAD 12.5 mg; QR-010 SAD 25 mg; QR-010 SAD 50 mg: QR-010 administered via inhalation as a single dose. QR-010: Single-stranded RNA antisense oligonucleotide in aqueous solution for oral inhalation
- Placebo SAD: Placebo (normal saline) administered via inhalation as a single dose Placebo: Normal Saline
- QR-010 MAD 6.25; QR-010 MAD 12.5 mg; QR-010 MAD 25 mg; QR-010 MAD 50 mg: QR-010 administered via inhalation three times weekly for four weeks. QR-010: Single-stranded RNA antisense oligonucleotide in aqueous solution for oral inhalation.
- Placebo MAD: Placebo (normal saline) administered via inhalation three times weekly for four weeks.
  Placebo: Normal Saline
Period: Single Ascending Dose (SAD) Cohorts
Arm/Group | QR-010 SAD 6.25mg | QR-010 SAD 12.5 mg | QR-010 SAD 25 mg | QR-010 SAD 50 mg | Placebo SAD | QR-010 MAD 6.25 | QR-010 MAD 12.5 mg | QR-010 MAD 25 mg | QR-010 MAD 50 mg | Placebo MAD
Started | 6 | 6 | 9 | 6 | 9 | 0 | 0 | 0 | 0 | 0
Completed | 6 | 6 | 9 | 6 | 9 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Multiple Ascending Dose (MAD) Cohorst
Arm/Group | QR-010 SAD 6.25mg | QR-010 SAD 12.5 mg | QR-010 SAD 25 mg | QR-010 SAD 50 mg | Placebo SAD | QR-010 MAD 6.25 | QR-010 MAD 12.5 mg | QR-010 MAD 25 mg | QR-010 MAD 50 mg | Placebo MAD
Started | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 7 | 6 | 9
Completed | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 5 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Met stopping criteria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- QR-010 SAD 6.25 mg; QR-010 SAD 12.5 mg; QR-010 SAD 25 mg; QR-010 SAD 50 mg: QR-010 administered via inhalation as a single dose
  QR-010: Single-stranded RNA antisense oligonucleotide in aqueous solution for oral inhalaton
- QR-010 MAD 6.25 mg; QR-010 MAD 12.5 mg; QR-010 MAD 25 mg; QR-010 MAD 50 mg: QR-010 administered via inhalation three times weekly for four weeks.
  QR-010: Single-stranded RNA antisense oligonucleotide in aqueous solution for oral inhalaton
- Total: Total of all reporting groups
Arm/Group | QR-010 SAD 6.25 mg | QR-010 SAD 12.5 mg | QR-010 SAD 25 mg | QR-010 SAD 50 mg | Placebo SAD | QR-010 MAD 6.25 mg | QR-010 MAD 12.5 mg | QR-010 MAD 25 mg | QR-010 MAD 50 mg | Placebo MAD | Total
Number analyzed (Participants) | 6 | 6 | 9 | 6 | 9 | 6 | 6 | 7 | 6 | 9 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 9 | 6 | 9 | 6 | 6 | 7 | 6 | 9 | 70
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.8 (8.01) | 21.5 (2.95) | 27.2 (7.31) | 22.7 (3.88) | 24.8 (8.26) | 22.7 (2.66) | 27.7 (10.42) | 32.3 (10.63) | 23.3 (4.18) | 26.3 (6.69) | 25.6 (7.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 5 | 2 | 3 | 3 | 3 | 5 | 2 | 6 | 38
  Male | 2 | 1 | 4 | 4 | 6 | 3 | 3 | 2 | 4 | 3 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 6 | 9 | 6 | 9 | 6 | 6 | 7 | 6 | 9 | 70
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
  Belgium | 1 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 2 | 9
  United States | 1 | 1 | 4 | 5 | 1 | 1 | 1 | 0 | 1 | 3 | 18
  Czechia | 2 | 2 | 0 | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 9
  Denmark | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 2 | 1 | 1 | 8
  Italy | 1 | 1 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 7
  United Kingdom | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 3 | 8
  France | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Germany | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 6
Weight (kg) [Mean (Standard Deviation); unit: kg] | 59.4 (9.28) | 64.8 (2.26) | 67.5 (13.00) | 57.7 (9.70) | 62.2 (6.48) | 66.8 (6.87) | 62.6 (8.97) | 67.1 (4.35) | 61.3 (13.37) | 59.6 (9.19) | 63.0 (9.11)
BMI [Mean (Standard Deviation); unit: kg/m2] | 22.1 (2.54) | 24.1 (2.33) | 23.0 (2.59) | 21.5 (2.91) | 21.4 (1.73) | 23.5 (2.76) | 22.8 (2.65) | 23.6 (1.56) | 21.3 (2.86) | 20.9 (1.56) | 22.3 (2.42)
FEV1 [Mean (Standard Deviation); unit: L] — Lung function; forced expiratory volume in 1 second
  L | 3.24 (0.877) | 3.15 (0.666) | 3.78 (1.092) | 3.06 (0.700) | 3.64 (0.748) | 3.49 (0.590) | 3.19 (0.600) | 2.85 (0.577) | 3.40 (0.993) | 3.18 (0.778) | 3.32 (0.792)
ppFEV1 [Mean (Standard Deviation); unit: percent] — Lung function; percent predicted Forced Expiratory Volume in 1 second
  percent | 92.3 (13.31) | 91.4 (19.93) | 97.3 (20.39) | 80.9 (8.99) | 91.8 (12.91) | 90.7 (14.28) | 89.0 (14.21) | 79.9 (10.14) | 84.7 (13.59) | 86.7 (11.91) | 88.8 (14.54)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Subjects Experiencing Treatment Emergent Adverse Events From Baseline Through End of Study
Description: Number of subjects experiencing at least one treatment emergent adverse events (TEAEs)
Time Frame: 8 Days for Single-dose cohorts; 8 weeks for Multiple-dose cohorts
Population: All subjects who received either QR-010 or placebo
Measure: Count of Participants; unit: Participants
Arm/Group | QR-010 SAD 6.25 mg | QR-010 SAD 12.5 mg | QR-010 SAD 25 mg | QR-010 SAD 50 mg | Placebo SAD | QR-010 MAD 6.25 mg | QR-010 MAD 12.5 mg | QR-010 MAD 25 mg | QR-010 MAD 50 mg | Placebo MAD
Number analyzed (Participants) | 6 | 6 | 9 | 6 | 9 | 6 | 6 | 7 | 6 | 9
Participants | 3 | 2 | 7 | 4 | 2 | 5 | 5 | 6 | 5 | 9

2. Primary Outcome: Severity of Treatment Emergent Adverse Events From Baseline Through End of Study
Description: Assessment of severity of treatment emergent adverse events (TEAEs).
  Severity is graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events Modified for CF (CTCAE v4.03). For events not present in this listing the following grading was applied:
  Mild: Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated; Moderate: Minimal, local, or noninvasive intervention indicated; discomfort sufficient to reduce or interfere with daily activities; Severe: Medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization may be indicated; disabling; limits self-care with significant interference with daily activities; incapacitating with inability to perform self care activities of daily living; Life-threatening: Urgent intervention indicated; immediate risk of death.
Time Frame: 8 Days for Single-dose cohorts; 8 weeks for Multiple-dose cohorts
Population: All subjects who received either QR-010 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | QR-010 SAD 6.25 mg | QR-010 SAD 12.5 mg | QR-010 SAD 25 mg | QR-010 SAD 50 mg | Placebo SAD | QR-010 MAD 6.25 mg | QR-010 MAD 12.5 mg | QR-010 MAD 25 mg | QR-010 MAD 50 mg | Placebo MAD
Number analyzed (Participants) | 6 | 6 | 9 | 6 | 9 | 6 | 6 | 7 | 6 | 9
Participants
  Mild | 3 | 2 | 5 | 4 | 2 | 5 | 4 | 5 | 1 | 5
  Moderate | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 4 | 3
  Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Life-Threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Incidence of Subjects Experiencing Dose-Limiting Toxicities (DLT) in Each Dose Cohort From Baseline Through End of Study Visit.
Description: DLT's were defined as an allergic reaction, acute bronchospasm or acute AEs of interest requiring (immediate) medical intervention.
Time Frame: 8 Days for Single-dose cohorts; 8 weeks for Multiple-dose cohorts
Population: All subjects who received either QR-010 or placebo. There were no Dose Limiting Toxicities (DLTs) reported in the SAD or MAD cohorts.
Measure: Count of Participants; unit: Participants
Arm/Group | QR-010 SAD 6.25 mg | QR-010 SAD 12.5 mg | QR-010 SAD 25 mg | QR-010 SAD 50 mg | Placebo SAD | QR-010 MAD 6.25 mg | QR-010 MAD 12.5 mg | QR-010 MAD 25 mg | QR-010 MAD 50 mg | Placebo MAD
Number analyzed (Participants) | 6 | 6 | 9 | 6 | 9 | 6 | 6 | 7 | 6 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Subjects With Abnormalities Reported Regarding Laboratory Parameters, Vital Signs, ECG, Spirometry, and Physical Findings.
Description: Number of subjects experiencing at least one abnormality for the categories laboratory parameters, vital signs, ECG, spirometry and physical findings that were reported as treatment emergent adverse event with a relationship to study drug as either possibly, probably or definitely.
Time Frame: 8 Days for Single-dose cohorts; 8 weeks for Multiple-dose cohorts
Population: All subjects who received either QR-010 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | QR-010 SAD 6.25 mg | QR-010 SAD 12.5 mg | QR-010 SAD 25 mg | QR-010 SAD 50 mg | Placebo SAD | QR-010 MAD 6.25 mg | QR-010 MAD 12.5 mg | QR-010 MAD 25 mg | QR-010 MAD 50 mg | Placebo MAD
Number analyzed (Participants) | 6 | 6 | 9 | 6 | 9 | 6 | 6 | 7 | 6 | 9
Participants
  laboratory parameters | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
  vital signs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ECG | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Spirometry | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
  physical findings | 2 | 2 | 2 | 3 | 0 | 3 | 4 | 1 | 1 | 4

5. Secondary Outcome: Maximum Serum Concentration
Description: Cmax: QR-010 maximum serum concentrations
Time Frame: 8 Days for Single-dose cohorts; 8 weeks for Multiple-dose cohorts
Population: Study population included all subjects treated either with QR-010 or placebo. Quantifiable serum concentrations are only available for the 50mg SAD and 50 mg MAD cohorts.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | QR-010 SAD 6.25 mg | QR-010 SAD 12.5 mg | QR-010 SAD 25 mg | QR-010 SAD 50 mg | Placebo SAD | QR-010 MAD 6.25 mg | QR-010 MAD 12.5 mg | QR-010 MAD 25 mg | QR-010 MAD 50 mg | Placebo MAD
Number analyzed (Participants) | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 6 | 0
ng/mL
  Dose 1 |  |  |  | 2.9 (1.2) |  |  |  |  | 4.53 (3.38) |
  Week 4, Dose 12 |  |  |  | NA (NA) — for SAD cohorts, there is no Week 4, Dose 12 timepoint |  |  |  |  | 3.63 (2.73) |

6. Secondary Outcome: Time to Maximum Serum Concentration
Description: Tmax: Time to Cmax of QR-010 serum concentrations.
Time Frame: 8 Days for Single-dose cohorts; 8 weeks for Multiple-dose cohorts
Population: Population included all subjects treated with either QR-010 or placebo. Quantifiable serum concentrations are only available for the 50mg SAD and MAD cohorts.
Measure: Median (Full Range); unit: hour
Arm/Group | QR-010 SAD 6.25 mg | QR-010 SAD 12.5 mg | QR-010 SAD 25 mg | QR-010 SAD 50 mg | Placebo SAD | QR-010 MAD 6.25 mg | QR-010 MAD 12.5 mg | QR-010 MAD 25 mg | QR-010 MAD 50 mg | Placebo MAD
Number analyzed (Participants) | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 6 | 0
hour
  Dose 1 |  |  |  | 0.6 [0.5 to 2.1] |  |  |  |  | 0.5 [0.5 to 3.0] |
  Week 4, Dose 12 |  |  |  | NA [NA to NA] — for SAD cohorts, there is no Week 4, Dose 12 timepoint |  |  |  |  | 1.0 [1.0 to 2.0] |

7. Secondary Outcome: Terminal Half-life (T1/2)
Description: The terminal elimination half-life will be estimated by non-linear regression analysis of the terminal elimination slope
Time Frame: 8 Days for Single-dose cohorts; 8 weeks for Multiple-dose cohorts
Population: The terminal half-life is not reported because the %AUC (Area Under the Curve) extrapolation was too large.
Arm/Group | QR-010 SAD 6.25 mg | QR-010 SAD 12.5 mg | QR-010 SAD 25 mg | QR-010 SAD 50 mg | Placebo SAD | QR-010 MAD 6.25 mg | QR-010 MAD 12.5 mg | QR-010 MAD 25 mg | QR-010 MAD 50 mg | Placebo MAD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Area Under the Curve to Final Sample [AUC(0-last)]
Description: Area under the curve to the final sample with a concentration greater than lower limit of quantification (LLQ) will be calculated using the linear trapezoidal method
Time Frame: 8 Days for Single-dose cohorts; 8 weeks for Multiple-dose cohorts
Population: Quantifiable serum concentrations are only available for the 50mg SAD and MAD cohort. For the PK parameters of the SAD 6.25, 12.5 and 25mg cohorts, no quantifiable serum concentrations could be measured. For the 6.25, 12.5 and 25mg MAD cohorts, no PK profiling was performed due to the large number of samples below the limit of detection.
Measure: Mean (Standard Deviation); unit: ng.hr/mL
Arm/Group | QR-010 SAD 6.25 mg | QR-010 SAD 12.5 mg | QR-010 SAD 25 mg | QR-010 SAD 50 mg | Placebo SAD | QR-010 MAD 6.25 mg | QR-010 MAD 12.5 mg | QR-010 MAD 25 mg | QR-010 MAD 50 mg | Placebo MAD
Number analyzed (Participants) | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 6 | 0
ng.hr/mL
  Dose 1 |  |  |  | 17.2 (8.2) |  |  |  |  | 19.0 (15.6) |
  Week 4, Dose 12 |  |  |  | NA (NA) — for SAD cohorts, there is no Week 4, Dose 12 timepoint |  |  |  |  | 17.0 (11.4) |

9. Secondary Outcome: Area Under the Curve to Infinity [AUC(0-∞)]
Description: AUC0-∞: Area under the curve to infinity will be calculated based on the last observed concentration Clast(obs) using formula: AUC0-∞=AUClast+Clast(obs)/λz
Time Frame: 8 Days for Single-dose cohorts; 8 weeks for Multiple-dose cohorts
Population: The Area Under the Curve to Infinity is not reported because the %AUC extrapolation was too large
Arm/Group | QR-010 SAD 6.25 mg | QR-010 SAD 12.5 mg | QR-010 SAD 25 mg | QR-010 SAD 50 mg | Placebo SAD | QR-010 MAD 6.25 mg | QR-010 MAD 12.5 mg | QR-010 MAD 25 mg | QR-010 MAD 50 mg | Placebo MAD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Serum Clearance (CL)
Description: CL: Serum clearance will be estimated using the formula: CL = Dose/AUC0-∞.
Time Frame: 8 Days for Single-dose cohorts; 8 weeks for Multiple-dose cohorts
Population: The Serum Clearance is not reported because the %AUC extrapolation was too large.
Arm/Group | QR-010 SAD 6.25 mg | QR-010 SAD 12.5 mg | QR-010 SAD 25 mg | QR-010 SAD 50 mg | Placebo SAD | QR-010 MAD 6.25 mg | QR-010 MAD 12.5 mg | QR-010 MAD 25 mg | QR-010 MAD 50 mg | Placebo MAD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Other Pre Specified Outcome: Adjusted Mean Change From Baseline in CFQ-R RSS
Description: Patient Reported Outcome measure Cystic Fibrosis Questionnaire-Revised Respiratory Symptom Score (CFQ-R RSS). A higher score represents a better outcome. A minimal clinically important difference (MCID) in the respiratory domain (CFQ-R RSS) has been established in stable populations as 4.0 points, and a maximum score is 100 points. Mean values reported refer to ''adjusted mean change from baseline'' values.
Time Frame: Day 15, Day 33, Day 54
Population: All subjects treated with either QR-010 or placebo in the Multiple Ascending Dose cohorts that received at least 10 out of 12 doses.
  For 1 subject in the placebo group no data were available at Day 54. "Mean" in this table refers to "Adjusted Mean".
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | QR-010 MAD 6.25 mg | QR-010 MAD 12.5 mg | QR-010 MAD 25 mg | QR-010 MAD 50 mg | Placebo MAD
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 8
score on a scale
  Day 15 | -4.13 (4.10) | 8.95 (4.12) | 7.76 (4.15) | -0.80 (4.51) | -5.09 (3.59)
  Day 33 | 6.43 (4.92) | 12.65 (4.93) | 7.76 (4.96) | -3.02 (5.40) | -6.48 (4.29)
  Day 54: number analyzed (Participants) | 6 | 6 | 6 | 5 | 7
  Day 54 | -10.24 (6.56) | 0.61 (6.57) | 5.91 (6.59) | -4.13 (7.20) | -10.31 (5.87)

12. Other Pre Specified Outcome: Adjusted Mean Change From Baseline in CFQ-R RSS as Compared to Placebo
Description: as for outcome 11
Time Frame: Day 15, Day 33, Day 54
Population: All subjects treated with either QR-010 or placebo in the Multiple Ascending Dose cohorts that received at least 10 out of 12 doses.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | QR-010 MAD 6.25 mg | QR-010 MAD 12.5 mg | QR-010 MAD 25 mg | QR-010 MAD 50 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5
score on a scale
  Day 15 | 0.96 (5.46) | 14.03 (5.49) | 12.85 (5.55) | 4.29 (5.73)
  Day 33 | 12.91 (6.53) | 19.13 (6.56) | 14.24 (6.60) | 3.46 (6.87)
  Day 54 | 0.07 (8.81) | 10.92 (8.83) | 16.22 (8.87) | 6.18 (9.26)
Statistical Analysis 1: Comparison: QR-010 MAD 6.25 mg; A mixed-model analysis was performed with repeated time measures on the change from baseline CFQ-R RSS as outcome variable and including treatment, baseline CFQ-R RSS value, time and interaction between time and treatment as covariates; Test type: Superiority; p = 0.0592, Mixed Models Analysis — p-values are presented for Day 33; Difference vs placebo = 12.91, 95% CI 2-sided [-0.54 to 26.35], Standard Error of Mean 6.53
Statistical Analysis 2: Comparison: QR-010 MAD 12.5 mg; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.0074, Mixed Models Analysis — p-values are presented for Day 33; difference vs placebo = 19.13, 95% CI 2-sided [5.62 to 32.64], Standard Error of Mean 6.56
Statistical Analysis 3: Comparison: QR-010 MAD 25 mg; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.0408, Mixed Models Analysis — p-values are presented for Day 33; difference vs placebo = 14.24, 95% CI 2-sided [0.64 to 27.83], Standard Error of Mean 6.60
Statistical Analysis 4: Comparison: QR-010 MAD 50 mg; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.6193, Mixed Models Analysis — p-values are presented for Day 33; difference vs placebo = 3.46, 95% CI 2-sided [-10.69 to 17.60], Standard Error of Mean 6.87

13. Other Pre Specified Outcome: Adjusted Mean Change From Baseline in CFQ-R RSS (Subgroup ppFEV1 <90% at Baseline)
Description: as for outcome 11
Time Frame: Day 15, Day 33, Day 54
Population: Subjects treated with either QR-010 or placebo in the Multiple Ascending Dose cohorts that received at least 10 out of 12 doses, with ppFEV1 <90% at baseline.
  For 1 subject in the placebo group no data were available at Day 54. "Mean" in this table refers to "Adjusted Mean".
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | QR-010 MAD 6.25 mg | QR-010 MAD 12.5 mg | QR-010 MAD 25 mg | QR-010 MAD 50 mg | Placebo MAD
Number analyzed (Participants) | 3 | 4 | 5 | 4 | 4
score on a scale
  Day 15 | -3.37 (5.51) | 8.64 (4.87) | 9.56 (4.28) | -0.87 (4.79) | -4.77 (4.82)
  Day 33 | 11.45 (7.36) | 15.58 (6.44) | 8.44 (5.71) | -0.87 (6.38) | -11.72 (6.41)
  Day 54: number analyzed (Participants) | 3 | 4 | 5 | 4 | 3
  Day 54 | -3.37 (6.36) | 5.86 (5.59) | 7.33 (4.94) | -3.65 (5.52) | -6.49 (6.33)

14. Other Pre Specified Outcome: Adjusted Mean Change From Baseline in CFQ-R RSS as Compared to Placebo (Subgroup ppFEV1 <90% at Baseline)
Description: Patient Reported Outcome measure Cystic Fibrosis Questionnaire-Revised Respiratory Symptom Score (CFQ-R RSS).
  A higher score represents a better outcome. A minimal clinically important difference (MCID) in the respiratory domain (CFQ-R RSS) has been established in stable populations as 4.0 points, and a maximum score is 100 points. Mean values reported refer to ''difference vs placebo in adjusted mean change from baseline'' values.
Time Frame: Day 15, Day 33, Day 54
Population: All subjects treated with either QR-010 or placebo in the Multiple Ascending Dose cohorts that received at least 10 out of 12 doses, with ppFEV1 <90% at Baseline.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | QR-010 MAD 6.25 mg | QR-010 MAD 12.5 mg | QR-010 MAD 25 mg | QR-010 MAD 50 mg
Number analyzed (Participants) | 3 | 4 | 5 | 4
score on a scale
  Day 15 | 1.41 (7.29) | 13.41 (6.95) | 14.33 (6.49) | 3.90 (6.74)
  Day 33 | 23.17 (9.73) | 27.30 (9.17) | 20.16 (8.62) | 10.84 (9.01)
  Day 54 | 3.12 (8.93) | 12.35 (8.58) | 13.82 (8.08) | 2.84 (8.33)
Statistical Analysis 1: Comparison: QR-010 MAD 6.25 mg; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.0321, Mixed Models Analysis — p-values are presented for Day 33; Difference vs placebo = 23.17, 95% CI 2-sided [2.29 to 44.04], Standard Error of Mean 9.73
Statistical Analysis 2: Comparison: QR-010 MAD 12.5 mg; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.0100, Mixed Models Analysis — p-values are presented for Day 33; Difference vs placebo = 27.30, 95% CI 2-sided [7.64 to 46.96], Standard Error of Mean 9.17
Statistical Analysis 3: Comparison: QR-010 MAD 25 mg; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.0346, Mixed Models Analysis — p-values are presented for Day 33; Difference vs placebo = 20.16, 95% CI 2-sided [1.68 to 38.64], Standard Error of Mean 8.62
Statistical Analysis 4: Comparison: QR-010 MAD 50 mg; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.2485, Mixed Models Analysis — p-values are presented for Day 33; Difference vs placebo = 10.84, 95% CI 2-sided [-8.47 to 30.16], Standard Error of Mean 9.01

15. Other Pre Specified Outcome: Adjusted Mean Change From Baseline in ppFEV1
Description: Exploratory efficacy parameter, as measured by spirometry, and expressed in percent predicted FEV1 (ppFEV1). Mean values reported refer to ''adjusted mean change from baseline'' values.
Time Frame: Day 15, Day 33, Day 54
Population: as for outcome 12
Measure: Mean (Standard Error); unit: percentage of predicted
Arm/Group | QR-010 MAD 6.25 mg | QR-010 MAD 12.5 mg | QR-010 MAD 25 mg | QR-010 MAD 50 mg | Placebo MAD
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 8
percentage of predicted
  (pre-dose) Day 15 | 0.06 (1.96) | 2.50 (1.96) | -4.03 (1.96) | -1.85 (2.14) | -0.83 (1.70)
  (pre-dose) Day 26 | 0.46 (2.64) | 3.22 (2.64) | -0.98 (2.64) | -1.39 (2.89) | -0.80 (2.28)
  Day 33 | 1.54 (2.40) | 0.05 (2.40) | -2.17 (2.40) | -3.21 (2.63) | -2.70 (2.08)
  Day 54 | 1.68 (2.88) | -1.63 (2.88) | 0.61 (2.88) | -2.43 (3.15) | -2.58 (2.49)

16. Other Pre Specified Outcome: Adjusted Mean Change From Baseline in ppFEV1 as Compared to Placebo
Description: Exploratory efficacy parameter, as measured by spirometry, and expresssed in percent predicted FEV1 (ppFEV1). Mean values reported refer to''difference vs placebo in adjusted mean change from baseline'' values.
Time Frame: Day 15, Day 33, Day 54
Population: as for outcome 12
Measure: Mean (Standard Error); unit: percentage of predicted
Arm/Group | QR-010 MAD 6.25 mg | QR-010 MAD 12.5 mg | QR-010 MAD 25 mg | QR-010 MAD 50 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5
percentage of predicted
  Day 15 | 0.89 (2.59) | 3.32 (2.59) | -3.20 (2.59) | -1.02 (2.73)
  Day 26 | 1.26 (3.49) | 4.02 (3.49) | -0.17 (3.49) | -0.59 (3.68)
  Day 33 | 4.24 (3.18) | 2.75 (3.18) | 0.53 (3.18) | -0.51 (3.35)
  Day 54 | 4.26 (3.81) | 0.96 (3.80) | 3.20 (3.81) | 0.15 (4.01)
Statistical Analysis 1: Comparison: QR-010 MAD 6.25 mg; A mixed-model analysis was performed with repeated time measures on the change from baseline ppFEV1 as outcome variable and including treatment, baseline ppFEV1 value, time and interaction between time and treatment as covariate; Test type: Superiority; p = 0.1938, Mixed Models Analysis — P-values are presented for Day 33; difference vs placebo = 4.24, 95% CI 2-sided [-2.30 to 10.79], Standard Error of Mean 3.18
Statistical Analysis 2: Comparison: QR-010 MAD 12.5 mg; A mixed-model analysis was performed with repeated time measures on the change from baseline ppFEV1 as outcome variable and including treatment, baseline ppFEV1 value, time and interaction between time and treatment as covariates; Test type: Superiority; p = 0.3943, Mixed Models Analysis — P-values are presented for Day 33; difference vs placebo = 2.75, 95% CI 2-sided [-3.79 to 9.29], Standard Error of Mean 3.18
Statistical Analysis 3: Comparison: QR-010 MAD 25 mg; [analysis description as in outcome 16, analysis 2]; Test type: Superiority; p = 0.8688, Mixed Models Analysis — P-values are presented for Day 33; difference vs placebo = 0.53, 95% CI 2-sided [-6.01 to 7.07], Standard Error of Mean 3.18
Statistical Analysis 4: Comparison: QR-010 MAD 50 mg; [analysis description as in outcome 16, analysis 2]; Test type: Superiority; p = 0.8813, Mixed Models Analysis — P-values are presented for Day 33; difference vs placebo = -0.51, 95% CI 2-sided [-7.41 to 6.39], Standard Error of Mean 3.35

17. Other Pre Specified Outcome: Adjusted Mean Change From Baseline in ppFEV1 (Subgroup ppFEV1 <90% at Baseline)
Description: Exploratory efficacy parameter, as measured by spirometry, and expresssed in percent predicted FEV1. Mean values reported refer to ''adjusted mean change from baseline'' values.
Time Frame: Day 15, Day 33, Day 54
Population: as for outcome 14
Measure: Mean (Standard Error); unit: percentage of predicted
Arm/Group | QR-010 MAD 6.25 mg | QR-010 MAD 12.5 mg | QR-010 MAD 25 mg | QR-010 MAD 50 mg | Placebo MAD
Number analyzed (Participants) | 3 | 4 | 5 | 4 | 4
percentage of predicted
  Day 15 | -0.29 (2.22) | 4.54 (1.92) | -3.45 (1.71) | -1.01 (1.91) | -3.40 (1.95)
  Day 26 | 4.21 (4.05) | 7.15 (3.51) | 0.89 (3.13) | -0.10 (3.50) | -3.76 (3.52)
  Day 33 | 6.01 (3.16) | 3.81 (2.74) | -0.68 (2.44) | -0.97 (2.73) | -4.18 (2.76)

18. Other Pre Specified Outcome: Adjusted Mean Change From Baseline in ppFEV1 as Compared to Placebo (Subgroup ppFEV1 <90% at Baseline)
Description: Exploratory efficacy parameter, as measured by spirometry, and expresssed in percent predicted FEV1. Mean values reported refer to ''difference vs placebo in adjusted mean change from baseline'' values.
Time Frame: Day 15, Day 33, Day 54
Population: Subjects treated with either QR-010 or placebo in the Multiple Ascending Dose cohorts that received at least 10 out of 12 doses, with ppFEV1 <90% at Baseline.
Measure: Mean (Standard Error); unit: percentage of predicted
Arm/Group | QR-010 MAD 6.25 mg | QR-010 MAD 12.5 mg | QR-010 MAD 25 mg | QR-010 MAD 50 mg
Number analyzed (Participants) | 3 | 4 | 5 | 4
percentage of predicted
  Day 15 | 3.11 (2.99) | 7.93 (2.76) | -0.05 (2.59) | 2.38 (2.74)
  Day 26 | 7.97 (5.39) | 10.90 (4.98) | 4.65 (4.71) | 3.65 (4.97)
  Day 33 | 10.19 (4.22) | 7.99 (3.91) | 3.50 (3.69) | 3.21 (3.89)
Statistical Analysis 1: Comparison: QR-010 MAD 6.25 mg; Test type: Superiority; p = 0.0301, Mixed Models Analysis — P-values are presented for Day 33; Difference vs placebo = 10.19, 95% CI 2-sided [1.13 to 19.25], Standard Error of Mean 4.22
Statistical Analysis 2: Comparison: QR-010 MAD 12.5 mg; Test type: Superiority; p = 0.0601, Mixed Models Analysis — P-values are presented for Day 33; Difference vs placebo = 7.99, 95% CI 2-sided [-0.39 to 16.37], Standard Error of Mean 3.91
Statistical Analysis 3: Comparison: QR-010 MAD 25 mg; Test type: Superiority; p = 0.3580, Mixed Models Analysis — P-values are presented for Day 33; Difference vs placebo = 3.50, 95% CI 2-sided [-4.40 to 11.41], Standard Error of Mean 3.69
Statistical Analysis 4: Comparison: QR-010 MAD 50 mg; Test type: Superiority; p = 0.4224, Mixed Models Analysis — P-values are presented for Day 33; Difference vs placebo = 3.21, 95% CI 2-sided [-5.13 to 11.55], Standard Error of Mean 3.89

ADVERSE EVENTS:
Time Frame: For the SAD cohorts, from randomization up to Day 8 after dose administration. For the MAD cohorts, from randomization for at least 30 days after the last administration of the study treatment.
Arm/Group | QR-010 SAD 6.25 mg | QR-010 SAD 12.5 mg | QR-010 SAD 25 mg | QR-010 SAD 50 mg | Placebo SAD | QR-010 MAD 6.25 mg | QR-010 MAD 12.5 mg | QR-010 MAD 25 mg | QR-010 MAD 50 mg | Placebo MAD
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/9 | 0/6 | 0/9 | 0/6 | 0/6 | 0/7 | 0/6 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/9 | 0/6 | 0/9 | 0/6 | 0/6 | 0/7 | 1/6 | 1/9
Other Adverse Events (participants affected / at risk) | 3/6 | 2/6 | 7/9 | 4/6 | 2/9 | 5/6 | 5/6 | 6/7 | 5/6 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | QR-010 SAD 6.25 mg (N=6) | QR-010 SAD 12.5 mg (N=6) | QR-010 SAD 25 mg (N=9) | QR-010 SAD 50 mg (N=6) | Placebo SAD (N=9) | QR-010 MAD 6.25 mg (N=6) | QR-010 MAD 12.5 mg (N=6) | QR-010 MAD 25 mg (N=7) | QR-010 MAD 50 mg (N=6) | Placebo MAD (N=9)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Calculus Urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QR-010 SAD 6.25 mg (N=6) | QR-010 SAD 12.5 mg (N=6) | QR-010 SAD 25 mg (N=9) | QR-010 SAD 50 mg (N=6) | Placebo SAD (N=9) | QR-010 MAD 6.25 mg (N=6) | QR-010 MAD 12.5 mg (N=6) | QR-010 MAD 25 mg (N=7) | QR-010 MAD 50 mg (N=6) | Placebo MAD (N=9)
Headache (Nervous system disorders) | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Forced expiratory volume decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 3 | 1 | 0 | 2 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 — General disorders and administration site conditions
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 — General disorders and administration site conditions

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators are restricted from disclosure or results until after multicenter publication or 12 months after the completion of the Study at all participating research centers. Sponsor can review results communication prior to public release and can embargo communications regarding trial results for a period that is more than 45 days (varying per site). Sponsor may request redaction of confidential information.

DOCUMENTS (2):
  • Study Protocol (2017-04-04): https://cdn.clinicaltrials.gov/large-docs/64/NCT02532764/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT02532764/SAP_001.pdf